CLINICAL TRIAL: NCT03879447
Title: Observational Study on the Effectiveness and Safety of Integrative Korean Medicine Treatment for Patients With Low Back Pain or Sciatica Due to Lumbar Stenosis or Spondylolisthesis
Brief Title: Effectiveness and Safety of Korean Medicine for Low Back Pain or Sciatica Due to Lumbar Stenosis/Spondylolisthesis
Status: Active, not recruiting | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2018-09
Record Dates: First submitted 2019-03-05; First posted 2019-03-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Lumbar Spinal Stenosis; Lumbar Spondylolisthesis; Low Back Pain; Sciatica; Neurogenic Claudication
Keywords: Korean Medicine; Effectiveness; Numeric Rating Scale; Safety; Walking ability; Disability
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis; Low Back Pain; Sciatica | interventions — Phytotherapy; Bee Venoms; Acupuncture Therapy; Electroacupuncture; Cupping Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Lumbar stenosis group: Lumbar stenosis patients will be administered integrative Korean medicine treatment consisting of herbal medicine, Chuna manual medicine, bee venom pharmacopuncture and pharmacopuncture, acupuncture, electroacupuncture, cupping, and other interventions, as needed.
  Interventions: Drug: Herbal medicine; Procedure: Chuna manual medicine; Procedure: Bee venom pharmacopuncture; Procedure: Pharmacopuncture; Procedure: Acupuncture; Procedure: Electroacupuncture; Procedure: Cupping; Procedure: Other intervention(s)
- Lumbar spondylolisthesis group: Lumbar spondylolisthesis patients will be administered integrative Korean medicine treatment consisting of herbal medicine, Chuna manual medicine, bee venom pharmacopuncture and pharmacopuncture, acupuncture, electroacupuncture, cupping, and other interventions, as needed.
  Interventions: Drug: Herbal medicine; Procedure: Chuna manual medicine; Procedure: Bee venom pharmacopuncture; Procedure: Pharmacopuncture; Procedure: Acupuncture; Procedure: Electroacupuncture; Procedure: Cupping; Procedure: Other intervention(s)

INTERVENTIONS:
Drug: Herbal medicine — Herbal medicine will be administered in water-based decoction (120ml) and dried powder (2g) form (Ostericum koreanum, Eucommia ulmoides, Acanthopanax sessiliflorus, Achyranthes japonica, Psoralea corylifolia, Saposhnikovia divaricata, Cibotium barometz, Lycium chinense, Boschniakia rossica, Cuscuta chinensis, Glycine max, Atractylodes japonica) at the physician's discretion.
  Other Names: Traditional herbal medicine
Procedure: Chuna manual medicine — Chuna is a Korean manual therapy directed at the spine and joints that incorporates various spinal manual medicine techniques for joint mobilization involving high-velocity, low amplitude thrusts to joints slightly beyond the passive range of motion and gentle force to joints within the passive range of movement. Chuna manual medicine will be administered to the pelvic, lumbar, thoracic, and cervical vertebrae at the physician's discretion.
  Other Names: Chuna manipulation; Chuna spinal manipulation
Procedure: Bee venom pharmacopuncture — Bee venom pharmacopuncture will be administered only after confirming a negative response to hypersensitivity skin test. Diluted bee venom (saline:bee venom ratio, 10,000:1) filtered for allergens will usually be injected at 4-5 acupoints proximal to the dysfunctional site at the physician's discretion. Each acupuncture point will be injected to a total of 0.5-1 cc using disposable injection needles (CPL, 1 cc, 26G x 1.5 syringe, Shinchang medical co., Korea).
  Other Names: Bee venom acupuncture; Bee venom
Procedure: Pharmacopuncture — Pharmacopuncture consisting of select herbal ingredients will be administered at Hyeopcheok (Huatuo Jiaji, EX B2), Ah-shi points and local acupuncture points using disposable injection needles (CPL, 1 cc, 26G x 1.5 syringe, Shinchang medical co., Korea) at the physician's discretion.
Procedure: Acupuncture — Acupuncture treatment will be administered using mainly proximal acupuncture points and Ah-shi points.
Procedure: Electroacupuncture — Electroacupuncture treatment will be administered using mainly proximal acupuncture points and Ah-shi points.
Procedure: Cupping — Cupping treatment will be administered at 1-2 points using mainly proximal acupuncture points and Ah-shi points.
Procedure: Other intervention(s) — Patients will be allowed any other additional intervention(s) as deemed necessary regardless of type or dose, and patterns of use will be investigated and recorded as a pragmatic clinical study.

SUMMARY:
A prospective observational study investigating the effectiveness and safety of integrative Korean medicine treatment in lumbar stenosis or spondylolisthesis patients with low back pain or sciatica at 3 locations of Jaseng Hospital of Korean Medicine as assessed through of pain, functional disability, walking ability, and quality of life patient-reported outcomes

DETAILED DESCRIPTION:
This is a prospective observational study to the aim of investigating the effectiveness and safety of integrative Korean medicine treatment (generally consisting of herbal medicine, Chuna manual medicine, bee venom pharmacopuncture and pharmacopuncture, acupuncture, electroacupuncture, and cupping) in lumbar stenosis or spondylolisthesis patients with low back pain or sciatica diagnosed by lumbar X-ray and/or MRI and clinical symptoms including neurogenic claudication at 3 locations of Jaseng Hospital of Korean Medicine (Bucheon, Daejeon, Busan (Haeundae)) as assessed through of pain, functional disability, walking ability, and quality of life patient-reported outcomes with a 5-year follow-up period

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiating leg pain or low back pain (LBP) intensity of NRS ≥5
* Patients diagnosed with lumbar stenosis based on dural sac cross-sectional area (DSCA) of <100 mm2 or morphological grading ≥B as assessed on MRI; or patients diagnosed with lumbar spondylolisthesis based on Meyerding Grade Ⅱ or higher as assessed on X-ray
* Clear neurogenic claudication symptoms (symptoms aggravated with walking, and alleviated upon resting in lumbar flexion position), if lumbar stenosis patient
* Patients with plans of receiving Korean medicine treatment for lumbar spinal stenosis for ≥4 months
* Patients who have agreed to study participation

Exclusion Criteria:

* Patients with vascular claudication
* Patients with other systemic diseases that may interfere with treatment effect or outcome interpretation
* Patients with soft tissue pathologies or pathologies of non-spinal origin that may cause LBP or radiating leg pain (e.g. spinal tumor, rheumatoid arthritis)
* Patients for whom acupuncture treatment may be inappropriate or unsafe (e.g. hemorrhagic diseases, blood clotting disorders, history of anti-coagulation medicine intake, serious diabetes with risk of infection, severe cardiovascular diseases, or other conditions deemed unsuitable for acupuncture treatment)
* Patients with medical history of spinal surgery within the past 3 months
* Patients who were treated with invasive interventions such as Korean medicine treatment, injections, physical therapy, or with medicine that may potentially influence pain such as NSAIDs (nonsteroidal antiinflammatory drugs) within the past week
* Pregnant patients or patients planning pregnancy
* Patients with serious psychological disorders
* Previous participation in other clinical studies within 1 month of current study enrollment, or plans to participate in other clinical studies during participation (including follow-up period) of the current study after study enrollment
* Patients unable to fill out study participation consent form
* Patients deemed unsuitable for study participation as assessed by the researchers

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lumbar stenosis or lumbar spondylolisthesis
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Numeric rating scale (NRS) of higher score at baseline out of low back pain or radiating leg pain | Change from baseline to 4 months
  Change from higher score at baseline out of low back pain or radiating leg pain intensity to same score at 4 months. Total score range: -10 (worse outcome) to 10 (better outcome)

SECONDARY OUTCOMES:
Numeric rating scale (NRS) of low back pain | Baseline, observation at least once a week for the duration of active treatment up to a maximum of 24 weeks (2, 4, 6, 8, 12, 16, 20, 24 weeks), 1, 3, 5 years
  Low back pain intensity for the past 3 days. Total score range: 0 (better outcome) to 10 (worse outcome)
Numeric rating scale (NRS) of radiating leg pain | Baseline, observation at least once a week for the duration of active treatment up to a maximum of 24 weeks (2, 4, 6, 8, 12, 16, 20, 24 weeks), 1, 3, 5 years
  Radiating leg pain intensity for the past 3 days. Total score range: 0 (better outcome) to 10 (worse outcome)
Visual analogue scale (VAS) of low back pain | Baseline, 2, 4, 6, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years
  Low back pain intensity for the past 3 days. Total score range: 0 (better outcome) to 100 (worse outcome)
Visual analogue scale (VAS) of radiating leg pain | Baseline, 2, 4, 6, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years
  Radiating leg pain intensity for the past 3 days. Total score range: 0 (better outcome) to 100 (worse outcome)
Oswestry Disability Index (ODI) | Baseline, 2, 4, 6, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years
  Functional disability questionnaire. The possible range of each item score is 0 to 5. Total score range: 0 (better outcome) to 100 (worse outcome)
Pain-free walking distance (average of the past 3 days) | Baseline, 2, 4, 6, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years
  Walking ability. Average pain-free walking distance during the past 3 days as recalled at each timepoint defined in Time Frame. Total score range: 0 (worse outcome) to no maximum limit (better outcome)
Maximum walking distance (average of the past 3 days) | Baseline, 2, 4, 6, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years
  Walking ability. Average maximum walking distance during the past 3 days as recalled at each timepoint defined in Time Frame. Total score range: 0 (worse outcome) to no maximum limit (better outcome)
Zurich Claudication Questionnaire | Baseline, 4, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years
  Claudication questionnaire. There are 12 questions for all patients, and a further 6 questions to measure treatment outcomes for those who have received treatment. The The Zurich Claudication Questionnaire consists of three subscales: (1) Symptom severity scale (items 1-7) which are subdivided into a pain domain (items 1-4) and a neuroischemic domain (items 5-7)]: The possible range of each item score is 1 to 5. (2) Physical function scale (items 8-12): The possible range of each item score is 1 to 4. (3) Patient satisfaction with treatment scale (questions 13-18): The possible range of each item score is 1 to 4. The result is expressed as a percentage of the maximum possible score. Total score range: 0% (better outcome) to 100% (worse outcome)
EuroQol 5-dimensions 5-levels (EQ-5D-5L) | Baseline, 2, 4, 6, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years
  Health-related quality of life questionnaire. Total score range: 11111 (better outcome) to 55555 (worse outcome)
Patient Global Impression of Change (PGIC) | 8, 16, 20, 24 weeks, 1, 3, 5 years
  Global patient-reported outcome. Total score range: 1 (better outcome) to 7 (worse outcome)
Use of other intervention(s) | Baseline, 2, 4, 6, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years
  Use of any other additional intervention(s) other than the integrative Korean medicine treatment administered by the attending physician (start date of treatment, end date of treatment, name of treatment, number of treatment sessions received, and other comments)
Physical examination | Baseline, 2, 4, 6, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years
  Lumbar physical examination
Adverse reaction | Baseline, every visit for the duration of active treatment up to a maximum of 24 weeks (2, 4, 6, 8, 12, 16, 20, 24 weeks), 1, 3, 5 years
  Safety
SF-36 | [Time Frame: Baseline, 4, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years]
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
EQ-VAS | Baseline, 2, 4, 6, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years
  The EQ VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'.

CONTACTS AND LOCATIONS:
Overall Officials: Sun-A Kim, KMD, Principal Investigator — Daejeon Jaseng Hospital of Korean Medicine; Hyun-Woo Cho, KMD, Principal Investigator — Haeundae Jaseng Hospital of Korean Medicine; Ji-Yun Seo, KMD, Principal Investigator — Bucheon Jaseng Hospital of Korean Medicine; Kyoung-Sun Park, KMD, Principal Investigator — Jaseng Hospital of Korean Medicine
Locations (1):
- Jaseng Medical Foundation, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No